CLINICAL TRIAL: NCT07338916
Title: Minimum Effective Volume (MEV90) of Local Anesthetic Required for Ultrasound-Guided Interscalene Block for Supraclavicular Nerve Block: A Dose-Finding Study
Brief Title: Dose-Finding Study: MEV90 for Local Anesthetic in Interscalene Block for Supraclavicular Nerves Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Trabajador de Santiago (Other)
Responsible Party: Principal Investigator, Germán Armando Aguilera Ceballos, Principal Investigator, Hospital del Trabajador de Santiago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Project Nº34, 2025; 251213001 (Other: Comité Ético Científico de Ciencias de la Salud - Universidad Católica)
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Brachial Plexus Blockade; Shoulder Surgery; Superficial Cervical Plexus Block
Keywords: Interscalene Block; Brachial Plexus Blockade; Supraclavicular nerves block; Shoulder Surgery; Miminum Effective Volume 90; MEV90
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minimum Effective Volume 90 (MEV90) (Experimental): Participants in this arm will receive a single-shot ultrasound-guided interscalene brachial plexus block as part of standard perioperative analgesia for shoulder arthroscopy. The intervention consists of injecting bupivacaine 0.5% with epinephrine (5 µg/mL) between the anterior and middle scalene muscles at the level of the C5-C6 nerve roots, using an in-plane technique under real-time ultrasound guidance.
  Interventions: Drug: Ultrasound-Guided Interscalene Block with Bupivacaine

INTERVENTIONS:
Drug: Ultrasound-Guided Interscalene Block with Bupivacaine — Participants will receive a single-shot interscalene brachial plexus block performed under real-time ultrasound guidance. The block targets the C5-C6 nerve roots between the anterior and middle scalene muscles using an in-plane technique. The local anesthetic is bupivacaine 0.5% with epinephrine (5 µg/mL). The injected volume ranges from 12 mL to 30 mL, determined by a dose-finding algorithm (biased coin up-and-down sequential design) to calculate the minimum effective volume (MEV90) for supraclavicular nerve block. All procedures are performed by experienced anesthesiologists following standard safety protocols, including incremental injection with aspiration and continuous monitoring (ECG, SpO₂, non-invasive blood pressure).

SUMMARY:
This study aims to determine the minimum effective volume (MEV90) of local anesthetic required to achieve sensory block of the supraclavicular nerves when performing a single-shot ultrasound-guided interscalene brachial plexus block (ISB). These nerves provide sensation to the skin over the clavicle and shoulder and are often involved in surgeries such as shoulder arthroscopy and clavicle repair.

DETAILED DESCRIPTION:
This prospective dose-finding study seeks to determine the minimum effective volume (MEV90) of local anesthetic required to achieve sensory block of the supraclavicular nerves following a single-shot ultrasound-guided interscalene brachial plexus block (ISB). These nerves, branches of the superficial cervical plexus, provide cutaneous innervation over the clavicle and shoulder and may contribute to postoperative pain after shoulder and clavicular surgery. Establishing MEV90 is clinically relevant to optimize analgesia while minimizing the risk of local anesthetic systemic toxicity.

The study employs a biased coin up-and-down sequential design, commonly used in regional anesthesia dose-finding trials. The initial volume is 12 mL of bupivacaine 0.5% with epinephrine (5 µg/mL), with subsequent volumes adjusted in 2 mL increments based on the prior patient's response. The maximum permitted volume is 30 mL.

All blocks are performed under ultrasound guidance by experienced anesthesiologists (≥60 ISBs), following standard safety protocols.

This intervention does not introduce additional risk beyond routine care, as ISB is the gold standard for shoulder surgery analgesia. Results will inform whether a single interscalene injection provides adequate coverage of supraclavicular nerves or if a separate cervical plexus block is necessary for procedures involving both plexuses, such as clavicle surgery. Findings may refine volume recommendations, improve analgesic strategies, and reduce unnecessary drug exposure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ASA physical status I to III
* Body Mass Index (BMI) between 18 and 35 kg/m²
* Weight ≥ 50 kg
* Scheduled for shoulder arthroscopy requiring an interscalene brachial plexus block for analgesia
* Able to provide informed consent

Exclusion Criteria:

* Inability to provide informed consent
* Coagulopathy (platelet count ≤100,000; INR ≥1.4)
* Significant pulmonary disease (restrictive or obstructive)
* Renal insufficiency (creatinine ≥1.2 mg/dL)
* Hepatic insufficiency (transaminases ≥100 U/L)
* Allergy to local anesthetics
* Pregnancy
* Pre-existing neuropathy
* Previous surgery in ipsilateral cervical or supraclavicular region
* Contralateral hemidiaphragmatic paralysis or vocal cord paralysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Minimum Effective Volume (MEV90) for Supraclavicular Nerve Block via Interscalene Approach | 30 minutes after completion of the block
  The primary outcome is the calculation of the minimum effective volume of local anesthetic (MEV90) required to achieve complete sensory block of the supraclavicular nerves following a single-shot ultrasound-guided interscalene brachial plexus block. Success is defined as absence of cold and touch sensation at the midpoint of the clavicle, assessed using an ice test.

SECONDARY OUTCOMES:
Sensorimotor Block Score for Interscalene Block | Every 5 minutes up to 30 minutes after block completion.
  Composite score (0-8 points) assessing sensory and motor block in C5-C6 dermatomes using ice test and motor function (shoulder abduction and external rotation). Success defined as ≥6 points.
Onset Time of Sensorimotor Block | Up to 30 minutes after block completion.
  Interval (minutes) between completion of local anesthetic injection and achievement of ≥6 points on the sensorimotor scale.
Sensory Block at Shoulder Arthroscopy Portals | 30 minutes after block completion.
  Presence or absence of cold and touch sensation at anterior, lateral, and posterior portal sites using ice test.
Sensory Block of Auricular, Occipital, and Transverse Cervical Nerves | 30 minutes after block completion.
  Assessment of sensory block in territories of auricular major, occipital minor, and transverse cervical nerves using ice test.
Pain Score During Block Procedure | Immediately after block completion.
  Patient-reported pain during needle insertion and injection, measured using Visual Analog Scale (VAS, 0-10).
Block Performance Times | During block procedure.
  Time intervals for image acquisition, needle placement, and total block execution (minutes).
Incidence of Block-Related Adverse Events | From block completion until end of surgery.
  Occurrence of complications including Horner's syndrome, hoarseness, dyspnea, vascular puncture, hematoma, paresthesia, and symptoms of local anesthetic systemic toxicity (LAST).

IPD SHARING:
Plan to Share IPD: No